CLINICAL TRIAL: NCT02134197
Title: An Open-label Phase I Dose-escalation Study to Evaluate the Safety, Tolerability, Maximum Tolerated Dose, Pharmacokinetics, and Pharmacodynamics of the Anti-C4.4a Antibody Drug Conjugate BAY1129980 in Subjects With Advanced Solid Tumors Known to Express C4.4a
Brief Title: Dose-escalation Study of Lupartumab Amadotin (BAY1129980)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16044
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Neoplasms
Keywords: Oncology; Solid tumors; Antibody drug conjugate; Maximum tolerated dose
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lupartumab Amadotin (BAY1129980) (Experimental): Dose escalation with consecutive expansion at MTD (maximum tolerated dose) with BAY1129980.
  Interventions: Drug: Lupartumab Amadotin (BAY1129980)

INTERVENTIONS:
Drug: Lupartumab Amadotin (BAY1129980) — Starting dose is 0.15mg/kg intravenous (I.V.) administration every 21 days.

SUMMARY:
The purpose of this study is to evaluate:

* The side effects of BAY1129980 when given every 21 days different dose levels.
* Determine the dose level of BAY1129980 that should be tested in future clinical research studies.
* Measure how much BAY1129980 is in the blood at specific times after administration.
* If treatment with BAY1129980 shows any effect on reducing the tumor growth.
* If there are specific biomarkers that might be able to explain why some patients respond to treatment and others do not.
* If treatment with BAY1129980 causes an immune response from the body against the drug (immunogenicity).

DETAILED DESCRIPTION:
The relatively restricted C4.4a expression pattern provides a target for the selective delivery of a cytotoxic drug to C4.4.a-expressing tumor cells by means of a suitable antibody-drug conjugate. The subject population eligible for the current study will be those subjects with advanced malignancies known to express C4.4a, which are refractory to standard therapy or those without standard therapy or actively refusing any treatment, which would be regarded as standard and in whom, in the opinion of the investigator, experimental therapy with BAY1129980 may be beneficial.Depending on the number of dose-escalating steps and the occurrence of DLTs, the planned numbers of subjects could vary.It is expected that up to 90 subjects may participate in the dose-expansion phase of the study and up to 6-9 subjects may particpate in the dose re-esclation phase.The study assessments in the expansion phase of the study are identical to those in the dose-escalation phase.

Amendment # 3 includes changes to DLT criteria (hematological and non-hematological) and allows for frequent follow-up for subjects experiencing drug-related liver toxicity that warrants dose reduction or dose interruptions.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be ≥ 18 years at the first screening examination / visit
* All subjects must provide a tumor tissue sample from [Formalin Fixed Paraffin Embedded (FFPE) slides] archival tissue or fresh biopsy collected before Cycle 1, Day 1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Life expectancy of at least 12 weeks
* Radiographically or clinically evaluable tumor. In the expansion phase, disease must be measurable according to RECIST 1.1.
* Adequate bone marrow, liver, and renal function
* Histologically or cytologically confirmed solid tumors known to express C4.4a (eg, carcinomas of the lung, head & neck SCC, esophagus SCC (squamous cell carcinoma),colon, ovary, prostate, and breast) that are refractory to any standard therapy, or have no standard therapy available, or for which subjects actively refuse any treatment that would be regarded as standard and in whom, in the opinion of the investigator, experimental therapy with BAY1129980 may be beneficial.
* A signed informed consent must be obtained prior to any study-specific procedures.
* Measurable disease with at least one lesion that can be accurately measured in at least one dimension according to RECIST 1.1

Exclusion Criteria:

* Anticancer chemotherapy, experimental cancer therapy, or cancer immunotherapy within 4 weeks prior to first dose study drug. Anticancer therapy is defined as any agent or combination of agents with clinically proven anti tumor activity administered by any route with the purpose of affecting the malignancy, either directly or indirectly, including palliative and therapeutic endpoints.
* Skin toxicity including but not limited to erythema, rash, ulceration, and open wound that is still clinically present and considered as acute or chronic.
* Subjects with psoriasis or other severe skin disease (eg, autoimmune skin disease, active erythematous skin lesions, etc.)
* Serious, non-healing wound, skin ulcer (of any grade), or bone fracture.
* Prior local radiotherapy is allowed if it is completed at least 4 weeks prior to the first dose of study drug and the subject has evaluable lesions not previously irradiated
* Significant liver dysfunction determined as Child-Pugh score B or C
* History of symptomatic metastatic brain or meningeal tumors unless the subject is >3 months from the end of definitive therapy before the first dose of study drug and has clinically or radiologically no evidence of tumor growth.
* History of clinically significant cardiac disease.
* Anti-platelet drugs within 4 weeks prior to the first dose of study drug. Anti-platelet drugs are defined as any agent or combination of agents with clinically proven anti-thrombotic activity administered by any route with the purpose of affecting blood clotting ability of the subject.
* Participation in another clinical trial in which they received active therapy within 4 weeks prior to the first dose of study drug.
* Subjects with CNS symptoms should undergo a CT scan or MRI of the brain to exclude new or progressive brain metastases. Spinal cord metastasis is acceptable. However, subjects with spinal cord compression should be excluded.
* Subjects with severe renal impairment (GFR <50 mL/min/1.73 m²) or on dialysis.
* History of organ allograft (except for corneal transplant) or autologous or allogeneic bone marrow transplant, or stem cell rescue within 3 months prior to the first dose of study drug.
* Current evidence or previous medical history of (ie, any absolute risk of latent infection) hepatitis B or C, any active hepatitis, or human immunodeficiency virus (HIV) infection. Active clinically serious infections > CTCAE Grade 2.
* Major surgery or significant trauma within 2 weeks prior to the first dose of study drug.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study result.
* Subjects who are pregnant or are breast-feeding.
* Any condition that is unstable or could jeopardize the safety of the subject and his / her compliance to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-05-22 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 21 days
  MTD is defined as the maximum dose at which the incidence of DLTs (dose limiting toxicities) during Cycle 1 is below 20%, or the maximum dose administered, whichever is achieved first during dose escalation.
Number of participants with adverse events as a measure of safety and tolerability | Up to 2 years

SECONDARY OUTCOMES:
C4.4a expression levels in tumour tissue as measured by immunohistochemistry (IHC) | Baseline
Tumor response evaluation following RECIST 1.1 criteria | Up to 2 years
Plasma concentration of BAY1129980 characterized by AUC (0-tlast) | 2 years
Antidrug and antibody titer | Baseline and up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- United States (15):
  - La Jolla, California
  - Stanford, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Georgia
  - Westwood, Kansas
  - Hackensack, New Jersey
  - Buffalo, New York
  - New York, New York
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Seattle, Washington

REFERENCES:
- [Derived] Willuda J, Linden L, Lerchen HG, Kopitz C, Stelte-Ludwig B, Pena C, Lange C, Golfier S, Kneip C, Carrigan PE, Mclean K, Schuhmacher J, von Ahsen O, Muller J, Dittmer F, Beier R, El Sheikh S, Tebbe J, Leder G, Apeler H, Jautelat R, Ziegelbauer K, Kreft B. Preclinical Antitumor Efficacy of BAY 1129980-a Novel Auristatin-Based Anti-C4.4A (LYPD3) Antibody-Drug Conjugate for the Treatment of Non-Small Cell Lung Cancer. Mol Cancer Ther. 2017 May;16(5):893-904. doi: 10.1158/1535-7163.MCT-16-0474. Epub 2017 Mar 14. PMID 28292941